CLINICAL TRIAL: NCT05996627
Title: Randomized Phase II Study of Belumosudil vs. Placebo for Preemptive Treatment of Chronic Graft Versus Host Disease
Brief Title: Belumosudil for the Pre-emptive Treatment of Patients With Chronic Graft Versus Host Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG1123523; NCI-2023-05293 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1123523 (Other: Fred Hutch/University of Washington Cancer Consortium); 20163 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil; KD025; Specimen Handling

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be conducted in a double-blinded fashion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Belumosudil) (Experimental): Patients receive belumosudil PO QD or BID if taken with strong CYP3A inducers or proton pump inhibitors for days 1 through 28 of each cycle. Cycles repeat every 28 days for a total of 11 cycles, followed by one cycle of tapering prior to discontinuation, in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection on study.
  Interventions: Drug: Belumosudil; Procedure: Biospecimen Collection; Other: Electronic Health Record Review
- Arm II (Placebo) (Placebo Comparator): Patients receive a placebo PO QD or BID if taken with strong CYP3A inducers or proton pump inhibitors for days 1 through 28 of each cycle. Cycles repeat every 28 days for a total of 11 cycles, followed by one cycle of tapering prior to discontinuation, in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Drug: Placebo Administration

INTERVENTIONS:
Drug: Belumosudil — Given PO
  Other Names: KD 025; KD-025; KD025; Rho-associated Coiled-coil Kinase 2 Inhibitor KD025; ROCK-II Inhibitor KD025; ROCK2 Inhibitor KD025; SLx 2119; SLx-2119; SLx2119
  Arms: Arm I (Belumosudil)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Ancillary studies
Drug: Placebo Administration — Given PO
  Arms: Arm II (Placebo)

SUMMARY:
This phase II trial compares the effect of belumosudil to a placebo in treating patients with chronic graft versus host disease. Chronic graft versus host disease remains a major complication of stem cell transplantation and can involve multiple organ systems. Belumosudil is a ROCK2 selective inhibitor that works to reduce the immune system response causing the chronic graft versus host disease. Giving belumosudil may better treat patients with chronic graft versus host disease and prevent the need for starting additional immune suppressive medications.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive belumosudil orally (PO) daily (QD) or twice daily (BID) if taken with strong CYP3A inducers or proton pump inhibitors for days 1 through 28 of each cycle. Cycles repeat every 28 days for a total of 11 cycles, followed by one cycle of tapering prior to discontinuation, in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive a placebo PO QD or BID if taken with strong CYP3A inducers or proton pump inhibitors for days 1 through 28 of each cycle. Cycles repeat every 28 days for a total of 11 cycles, followed by one cycle of tapering prior to discontinuation, in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection on study.

After completion of study treatment, patients are followed up at 30 days, at 60 days if 12 cycles are completed, and then up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* At least one diagnostic or distinctive cGVHD manifestation(s), with a clinical diagnosis of cGVHD,but patients do not need to meet National Institute of Health (NIH) criteria for cGVHD
* If eye involvement only, cGVHD must be confirmed on exam by an ophthalmologist or optometrist
* No new immune suppressive therapy added within preceding 2 weeks prior to study enrollment for any indication

  * Continuation of agents previously given as either GVHD prophylaxis or acute/late acute GVHD therapy are permitted. Modification of dose of these agents for targeting of therapeutic drug levels is permitted, as are decreases in existing prednisone or prednisone equivalent dose based on routine clinical tapering practices. Increases in prednisone or prednisone equivalents are not allowed in the 2 weeks prior to enrollment
* Age 18 and older
* Karnofsky performance score >= 70
* Able to take oral medications
* Signed informed consent
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN, unless due to Gilbert's disease
* Glomerular filtration rate (estimated glomerular filtration rate [eGFR]) >= 30 mL/min/1.73 m^2
* Female subjects of childbearing potential have a negative serum or urine pregnancy test at screening. Females of childbearing potential are defined as sexually mature females without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, females who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression
* Sexually active females of childbearing potential enrolled in the study must agree to use two forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes:

  * Intrauterine device (IUD) plus one barrier method
  * Stable doses of hormonal contraception for at least 3 months (eg, oral, injectable, implant, transdermal) plus one barrier method
  * 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gel that contain a chemical to kill sperm)
  * Surgical sterilization (tubal ligation)
  * A vasectomized partner
* For male subjects who are sexually active and who are partners of females of childbearing potential: Agreement to use two forms of contraception as per above and to not donate sperm during the treatment period and for at least 3 months after the last dose of study drug
* No evidence of active malignancy

Exclusion Criteria:

* Any systemic immune suppressive treatment for cGVHD (topical or local therapies are allowed)
* Plan to start systemic immune suppressive therapy for cGVHD or increase steroid dose within 14 days after planned start of study medication
* 0.25 mg/kg/day or higher prednisone or prednisone equivalent dose at time of screening
* History of non-compliance that in the investigator's opinion would interfere with study participation
* Uncontrolled psychiatric illness
* Female subject who is pregnant or breast feeding
* Previous therapy with belumosudil
* Known allergy/sensitivity to belumosudil or any other ROCK2 inhibitor
* Treatment with another investigational agent within 28 days (or 5 half-lives, whichever is greater) of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to start of subsequent systemic immune suppressive treatment for chronic graft versus host disease (cGVHD) | From first dose of study medication to starting a new systemic immunosuppressive agent for cGVHD therapy, up to 12 months
  Systemic therapies include any systemic agent given for a cGVHD indication, including extracorporeal photopheresis. Will use Gray's test. Point estimates of new systemic immunosuppressive use will be obtained using cumulative incidence estimates.

SECONDARY OUTCOMES:
Event-free survival | From randomization to death, malignancy relapse or addition of a new systemic immune suppressive therapy, up to 12 months or end of study
  Point estimates will be obtained using the method of Kaplan and Meier and the log-rank test will be used to assess the difference between treatment groups.
Overall survival | Up to 12 months or end of study
  Point estimates will be obtained using the method of Kaplan and Meier and the log-rank test will be used to assess the difference between treatment groups.
Rate of relapse | Up to 12 months or end of study
  Point estimates will be obtained using the method of Kaplan and Meier and the log-rank test will be used to assess the difference between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No